CLINICAL TRIAL: NCT04455880
Title: The Comparison of Placental Elastographic Values, Fetal and Neonatal Outcomes in Pregnant Women With Gestational Diabetes and Controls
Brief Title: Shear Wave Elastography in Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulsum Uysal (Other Government)
Responsible Party: Sponsor-Investigator, Gulsum Uysal, Associate Professor in Obstetrics and Gynecology Department, Adana Numune Training and Research Hospital
Organization: Adana Numune Training and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49/2019
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: Shear wave elastography; gestational diabetes mellitus; placental stiffness; high risk pregnancy; placenta
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Group 1 (n= 79, GDM with insulin therapy), Group 2 (n=90, GDM with only diet), Group 3 (n= 150, healthy controls) All patients were above 36 gestational weeks with anterior placenta.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GDM with insulin therapy (Active Comparator): Singleton pregnancies above 36 gestational weeks diagnosed Gestational Diabetes Mellitus and treated with insulin therapy.
  Interventions: Other: SWE is a novel noninvasive dynamic ultrasound technique which refers to measurement for quantitative analysis of tissue elasticity
- GDM treated with only diet (without any medical therapy) (Active Comparator): Singleton pregnancies above 36 gestational weeks diagnosed Gestational Diabetes Mellitus and treated with insulin therapy.
  Interventions: Other: SWE is a novel noninvasive dynamic ultrasound technique which refers to measurement for quantitative analysis of tissue elasticity
- Non-diabetic Controls (Active Comparator): Singleton non diabetic healthy pregnancies above 36 gestational weeks
  Interventions: Other: SWE is a novel noninvasive dynamic ultrasound technique which refers to measurement for quantitative analysis of tissue elasticity

INTERVENTIONS:
Other: SWE is a novel noninvasive dynamic ultrasound technique which refers to measurement for quantitative analysis of tissue elasticity — SWE is a novel noninvasive dynamic ultrasound technique which refers to measurement for quantitative analysis of tissue elasticity. The stiffer the tissue, the higher shear wave velocity is measured. Elastographic examinations were performed by physicians using Samsung HS70A ultrasound system with a Samsung CA1-7A convex transducer and S-Shear wave technique. During the examination, patients were lying in supine position, breathing levels kept steady to prevent noise and artifacts and minimum pressure were applied on the transducer to eliminate misleading tissue compression. A region of interest (ROI) box of 10 × 10 mm was positioned on placenta and six measurements were obtained from central and peripheral zones of placenta while avoiding vascular structures

SUMMARY:
Our aim was to investigate and compare placental elasticity by using Shear wave elastography (SWE) in patients with gestational diabetes mellitus (GDM) with and without insulin to non-diabetic controls.

This prospective study included 319 pregnant patients. Three groups were created as follows: Group 1 (n= 79, GDM with insulin therapy), Group 2 (n=90, GDM with only diet) and Group 3 (n= 150, healthy controls) All patients were above 36 gestational weeks with anterior placenta. Totally six measurements including the central and peripheral parts (right, left) of the placenta both from maternal and fetal sites were obtained with SWE. Demographic, obstetrics, fetal and perinatal features were also compared. Receiver operating characteristic analysis was plotted and cut-off of elastographic velocity values were noted

DETAILED DESCRIPTION:
This prospective study included singleton pregnant women aged between 18-45 years who applied for third trimester prenatal examination (36 gestational weeks and above) between May 2019 and December 2019 at Women and Children Disease Training and Research Hospital, Istanbul, Turkey. Ethical documents including Declaration of Helsinki were approved by local institutional review board (Approval number:49/2019) and a written informed consent was obtained from all patients. The study participants were divided into three groups according to treatments. While Group 1 consisted of patients with GDM using insulin therapy (GDM A2), patients with GDM treated with only diet (without any medical therapy) created Group 2 (GDM A1). Group 3 included healthy controls. Insulin therapy was initiated when target cut-off values were exceeded according to Carpenter and Coustan criteria. Patients with anterior placenta were included in the study because the effectiveness of the method decreased. Gestational age was recorded regarding last menstrual period and was checked in all participants by using a first trimester ultrasound report. All GDM patients were followed up in perinatology clinic and timing of delivery was organized individually basically on obstetrical indications. Ultrasonographic evaluation and SWE method were performed by single perinatologist Elastographic examinations were performed by physicians using Samsung HS70A ultrasound system with a Samsung CA1-7A convex transducer and S-Shear wave technique. During the examination, patients were lying in supine position, breathing levels kept steady to prevent noise and artifacts and minimum pressure were applied on the transducer to eliminate misleading tissue compression. A region of interest (ROI) box of 10 × 10 mm was positioned on placenta and six measurements were obtained from central and peripheral zones of placenta while avoiding vascular structures. Considering the disc-like structure of the placenta measurement areas were divided into six regions as follows: maternal right, maternal central, maternal left, fetal right, fetal central and fetal left. All measurements taken from different zones were recorded individually along with the mean value generated using IQR method. Through this approach, datasets were established not just for the auto-calculated mean value but also zone specific values for further analysis. All measurements were obtained in both kilopascal (kPa) and m/s formats.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnant women who applied for third trimester prenatal examination
* 36 gestational weeks and above with anterior placenta
* Diagnosed Gestational Diabetes Mellitus with 100 gr oral glucose tolerance test
* Using insulin therapy or diet without any anti-diabetic medication.

Exclusion Criteria:

* multiple gestations,
* pregnancies with fetal anomalies,
* morbidly adherent placenta and uterine malformations
* patients with systemic autoimmune diseases,
* patients with high blood pressure,
* patients with smoking history

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Singleton 36 weeks of gestation with anterior placenta
Enrollment: 319 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Shear wave elastography in gestational diabetes mellitus | 9 months
  To investigate and compare placental elasticity by using Shear wave elastography (SWE) in patients with gestational diabetes mellitus (GDM) with and without insulin to non-diabetic controls.
Prediction and differentiation of GDM and prognosis with Shear wave elastography velocity cut-offs | 9 months
  Cut off values of velocities will be estimated to predict GDM

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Acar Sirinoglu, MD, Principal Investigator — Zeynep Kamil Women and Children Disease Training and Research Hospital
Locations (1):
- Zeynep Kamil Women and Children Disease Training and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No